CLINICAL TRIAL: NCT04568252
Title: Evaluation of the Impact of Wearing a Millimetre Wave Bracelet for 3 Months on the Frequency in Number of Days of Migraines in Patients With Episodic Migraines Without Aura
Brief Title: Migraine STImulation Crisis of Migraine
Acronym: MISTIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Remedee SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MISTIC
Record Dates: First submitted 2020-07-31; First posted 2020-09-29 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Migraine Without Aura
Keywords: Migraine; Prophylaxis; Millimeter waves; Pain; Neuromodulation
MeSH Terms: conditions — Migraine without Aura; Migraine Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Randomization : intervention group and control group
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Millimetric wave emission bracelet.
  Interventions: Device: Wristband with millimeter wave emission.
- Control (Sham Comparator): Placebo bracelet.
  Interventions: Device: Placebo of wristband with millimeter wave emission.

INTERVENTIONS:
Device: Wristband with millimeter wave emission. — Wristband treatment with millimeter wave emission twice a day for 3 months.
  Arms: Intervention
Device: Placebo of wristband with millimeter wave emission. — Treatment with a millimeter wave emission wristband placebo twice a day for 3 months.
  Arms: Control

SUMMARY:
Migraine is a neurovascular disease whose prevalence is estimated at almost 20% of the adult population. Currently, there is no treatment for migraine.

Millimeter stimulation of the wrist subcutaneous receptors allows the release of endorphin in the brain.

MISTIC is a prospective, controlled, multicenter, double-blind, randomized study in which the research team are investigating whether millimeter stimulation of subcutaneous wrist receptors reduces the frequency of migraine crisis.

DETAILED DESCRIPTION:
MISTIC is a multicenter, controlled, randomized, double-blind study. Eligible patients will have to report their migraine crisis in a diary during a one month pre-selection phase. Then, patients will be randomized into one of two treatment groups :

* active millimeter wave emission bracelet
* or placebo bracelet

Patients will have to use the medical device twice a day for 3 months. The investigators will follow them for an additional 3 months to assess the persistence of the effect.

Throughout the follow-up, patients will report their migraines crisis in a journal.

The primary outcome will be the impact of wearing a millimeter wave bracelet for 3 months, on the number of days with migraine headaches.

ELIGIBILITY:
Inclusion Criteria:

* Patient with episodic migraine without aura (according to ICDH3 classification criteria)
* Patient with at leat 4 migraine days per month and no more than 8 migraine days per months
* Background treatment (or not) stable for at least 1 month
* Drug management of migraine stable for at least one month
* Non-drug management of stable migraine at least 1 month prior to the study
* Patient affiliated to social security or beneficiary of such a scheme

Exclusion Criteria:

* Patients with chronic migraine (defined according to IHS criteria)
* Patients already included in an interventional clinical research protocol
* Patients with chronic headache due to drug abuse (according to IHS criteria)
* Patients with only migraine crisis with aura
* Wrist size < 14.5 and > 21 cm
* Situations of dermatological pathologies on pre-existing wrists (oozing dermatosis, hyper sweating, eg.) or unhealed lesions on both wrists.
* Presence of metallic object (bracelet, watch, piercing...) on both wrists.
* Presence of a tattoo on both wrists
* Allergic reactions on contact with silicone or metal
* Persons referred to in Articles L 1121-5 to L 1121-8 of the CSP (corresponds to all protected persons) pregnant women, parturient women, nursing mothers, persons deprived of their liberty by judicial or administrative decision, persons subject to a legal protection measure
* Women of childbearing age with a short-term pregnancy project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of millimeter waves applied to the wrist (MMW) on the number of days with migraine(s) at 3 months reported by the patient with episodic migraine(s) without aura. | 3 months.
  Sequential hierarchical analysis on two criteria :
  * the difference in the number of days with migraine in the month prior to M3, taking into account the number of days with migraine in the month prior to inclusion, using an ANCOVA (comparison of average between the 2 groups adjusted to the initial value according to the recommendations of Vickers and Altman).
  * the difference in the proportion of success at M3 (reduction in the number of days with migraine by more than 50% between inclusion and M3), evaluated by the Chi2 test.

SECONDARY OUTCOMES:
To compare the evolution of migraine in terms of monthly monitoring. | 3 months.
  Comparison of the evolution's kinetic of the number of days with migraine between the baseline (M0) and 3 months using monthly data (M1-M2-M3).
To evaluate the effects of wearing a millimeter wave wristband on the severity of migraine crisis. | 3 months.
  Headache Impact Test (named HIT-6 questionnaire) Self-Rating Scale (3 levels : mild, moderate, severe).
  The HIT-6 questionnaire contains 6 questions (3 first questions assessing the impact of the crisis and 3 last questions assessing the impact of the crisis).
  The minimum score is 36 and the maximum score is 78. It can result in a categorical use to define four grades of increasing severity: score ≤ 49: low impact; score 50-50: definite impact; score 56-59: significant impact; score ≥ 60: impact major. The higher the score, the greater the impact of headaches on quality of life.
To evaluate the effects of wearing a millimeter wave wristband on the duration of migraine crisis. | 3 months.
  Duration (in minutes) of patient-reported migraine crisis at 3 months from baseline (M0).
Evaluation of the consumption of migraine crisis treatments between the 2 groups. | 3 months.
  Number of migraine crisis treatments.
To evaluate the effects of wearing the MMW wristband on the specific (i.e. migraine-related) quality of life of migraine patients (functional disability). | 3 months.
  Evolution of the MIDAS questionnaire score between 0 and M3. The MIDAS questionnaire contains 5 questions.
  Description of score : the higher the number of days, the higher severity :
  0 to 5 days : no severity 6 to 10 days : little severity 11 to 20 days : moderate severity more 20 days : high severity
To evaluate the effects of wearing the MMW wristband on generic quality of life. | 3 months.
  Evolution of the EQ5D-5L questionnaire score between 0 and M3. EQ-5D-5L is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of lige that can be used in a wide range of health conditions and treatments. The EQ5D has 6 items intended to measure general health. The top 5 rate mobility, independence, daily activities, pain / discomfort, and anxiety / depression, and are rated according to 5 values : "No problem", "little problem", "moderate problem", "high problem" and "Incapacity". This results in an index score. The last item deals with perceived health on the day the questionnaire is filled in and uses a visual analogue scale from 0 (wors) to 100 (best health possible) (Visual Analog Scale Score)
To evaluate the effects of wearing a millimeter wave wristband on associated anxiety and depressive disorders. | 3 months.
  Evolution of the HADS questionnaire between 0 and M3. The HADS questionnaire contains 14 questions. The minimum score is 0 and the maximum score is 42.
  The higher the score, the depression is important :
  score < 7 : no depression score 8 to 10 : doubtful depression score > 11 : proven depression
To evaluate the effects of wearing a millimeter wave wristband on the quality of sleep. | 3 months.
  Evolution of the MOS-Sleep questionnaire between 0 and M3. The PSQI questionnaire contains 12 questions. The minimum score is 0 and the maximum score is 100 : a score of 0 corresponds to a bad quality of spleep and a score of 100 to a good quality of spleep (no difficulties).
To evaluate the consumption in consultations (any type of care use) for migraine between the 2 groups. | 3 months.
  Comparison of the costs of consultations induced by migraine (hospitalizations, medical consultations).
To assess the consumption of complementary alternative migraine care between the 2 groups. | 3 months.
  Comparison of the number of complementary alternative consultations at 3 months between the 2 groups.
To evaluate the stability of the effect of wearing the MMW wristband over the long term in the intervention group. | 6 months.
  Evaluation of the maintenance of the stability of the effect of wearing the MMW at the long term (6 months) on the number of the migraine day for the principal outcome.
Adverse events. | 6 months.
  Description of adverse events from M0 to M6 (number and type)
To assess patient satisfaction with participation in the study. | 6 months.
  Questionnaire of satisfaction with the choice of treatment at 6 months. This questionnaire of satisfaction was created by our team in order to evaluate the satifaction of patient included in this study.
  It contains 13 questions. No score will be calculated, only description of answers.
Observance of the use of MMW wristband. | 3 months.
  Analysis of the recorded data related to the MMW wristband. The validation of the recordings is defined by the presence of at least 2/3 of the data during the total time of use of the bracelet during 3 months.
Subgroup analysis of the number of migraine day for the principal outcome in relation to patients with or without prior prophylactic treatment. | 6 months.
  To analyse if there is a best adaptation of treatment with ou without prior prophylactic treatment (stratification on the prior prophylactic treatment variable) on the number of migraine day for the principal outocme.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline MD MAINDET, Principal Investigator — CHUGA, 38000 Grenoble
Locations (6):
- France (6):
  - CHU Grenoble Alpes, Grenoble
  - Cabinet Mornant, Mornant
  - CH Fondation Rotschild, Paris
  - Cabinet Saint Ismier, Saint-Ismier
  - Cabinet Neuralpes, Saint-Martin-d'Hères
  - CH Voiron, Voiron